CLINICAL TRIAL: NCT06718829
Title: Effect of Core Stability and Sensorimotor Training Exercises on Postural Stability Post Lower Limb Burn
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rofaida Mohie Eldeen Ali Sobh, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/005151
Record Dates: First submitted 2024-12-02; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Burns
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Core Stability Exercises + Traditional physical therapy program (Experimental): This group will be composed of 30 patients with lower limb burns. Patients will receive core stability exercises in addition to a traditional physical therapy program in the form of stretching exercises, strengthening exercises and scar management. Exercises will be applied for 3 times a week for 8 consecutive weeks.
  Interventions: Other: Core Stability Exercises; Other: Traditional physical therapy program
- Sensorimotor Training Exercises + Traditional physical therapy program (Experimental): This group will be composed of 30 patients with lower limb burns. Patients will receive sensorimotor training exercise in addition to traditional physical therapy program in the form of stretching exercises, strengthening exercises and scar management. Exercises will be applied for 3 times a week for 8 consecutive weeks.
  Interventions: Other: Sensorimotor Training Exercises; Other: Traditional physical therapy program
- Core Stability Exercises + Sensorimotor Training Exercises + Traditional physical therapy program (Experimental): This group will be composed of 30 patients with lower limb burns. Patients will receive core stability exercises and sensorimotor training exercise in addition to traditional physical therapy program in the form of stretching exercises, strengthening exercises and scar management. Exercises will be applied for 3 times a week for 8 consecutive weeks.
  Interventions: Other: Core Stability Exercises; Other: Sensorimotor Training Exercises; Other: Traditional physical therapy program

INTERVENTIONS:
Other: Core Stability Exercises — Patients will perform core stability exercises three times weekly for eight weeks. The exercises include abdominal hollowing, bridge, right-angle leg lifts with thigh press, seated twist, knee-to-chest with elbow flexion, prone abdominal hollowing, prone arm and leg lift, quadruped abdominal hollowing, quadruped arm or arm-leg lifts, and various plank positions: forearm plank, side plank, forearm plank with hip raise, and forearm plank with straight legs.
  Arms: Core Stability Exercises + Sensorimotor Training Exercises + Traditional physical therapy program; Core Stability Exercises + Traditional physical therapy program
Other: Sensorimotor Training Exercises — Patients will perform sensorimotor training exercises three times weekly for eight weeks, progressing through three phases: static (weeks 1-2), dynamic (weeks 3-4), and functional (weeks 5-8). Exercises, repeated 3-5 times per session with rest intervals, advance from simple to complex as patients master each level. Static exercises include standing on firm/soft surfaces and single-leg balances. Dynamic exercises add forward lunges and T-band kicks. Functional training incorporates walking on various surfaces, toe and heel skipping, squats, balance drills on wobble boards, and multidirectional rolling movements with visual and single-leg variations. This progression enhances coordination, balance, and functional stability.
  Arms: Core Stability Exercises + Sensorimotor Training Exercises + Traditional physical therapy program; Sensorimotor Training Exercises + Traditional physical therapy program
Other: Traditional physical therapy program — All patients will undergo a traditional physical therapy program consisting of stretching exercises, strengthening exercises, and scar management techniques, three times weekly for eight weeks.

SUMMARY:
The purpose of the study is to determine the effect of core stability and sensorimotor training exercises on postural stability post lower limb burn.

DETAILED DESCRIPTION:
The need for this study develops from the lack of information in the published studies about the effectiveness of core stability exercises and sensorimotor training on the rehabilitation of burned patients.

Severe burn injuries, particularly those encompassing over 20% of the total body surface area (TBSA), trigger elevated catabolism and hypermetabolic responses in adult and pediatric burn patients. This wide spectrum of pronounced effects stemming from the hypermetabolic response and catabolism includes substantial muscle mass depletion, reduced muscle strength and endurance, hindered wound healing, impaired sensory perception, constrained ambulatory capacity, postural instability, and diminished functional mobility.

Core stability exercises improve neuromuscular system performance that causes the optimal lumbar-pelvic -hip chain mobility and good acceleration and deceleration, appropriate muscular balance, proximal stability and good function.

Sensorimotor training exercise emphasizes postural control and progressive challenges to the sensorimotor system to restore normal motor programs in patients. The proprio sensory system helps the motor system to maintain equilibrium on a reflex, automatic basis. In response to a sudden load, "the muscles will respond rapidly to stabilize the body, i.e., they will try to maintain balance and posture.

The present study is designed to investigate the effect of core stability and sensorimotor training exercises on postural stability in burned patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients are both males and females.
* Their age will range from (20-50) years.
* Patients will suffer from lower limb second degree burn (Partial thickness of thermal injury).
* Total body surface area (TBSA) for the burns will be ranged from 20% to 35% .
* Patients will begin the training program after complete wound healing.
* Patients will be given their informed consent.

Exclusion Criteria:

* Patients who had an open wound at or near treatment site.
* Patients who had chemical or electrical burn.
* Musculoskeletal disorders that will impair performance during training and tests.
* Uncontrolled cardiovascular or pulmonary diseases .
* Neurological and renal disorders.
* Metabolic or vascular disease with a neurological component such as diabetes.
* Malignant conditions.
* Psychiatric illness, severe behavior or cognitive disorders.
* Uncooperative patients.
* Pregnancy.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-12-10 (Estimated); Primary Completion 2025-05-10 (Estimated); Study Completion 2025-05-25 (Estimated)

PRIMARY OUTCOMES:
overall stability index | 8 weeks
  It was evaluated using the Biodex Balance System (BBS) before and after the eight-week treatment program. Patients will stand barefoot on the locked platform, centering themselves using visual feedback on the screen. Once stable, foot angles and heel coordinates will be recorded, and tests will commence with stability levels gradually decreasing from level eight to level four. Each test will last 30 seconds, with patients maintaining the cursor within the smallest balance zones. Postural stability measures will be calculated as the mean of three trials.
anterior-posterior stability index | 8 weeks
  It was evaluated using the Biodex Balance System (BBS) before and after the eight-week treatment program. Patients will stand barefoot on the locked platform, centering themselves using visual feedback on the screen. Once stable, foot angles and heel coordinates will be recorded, and tests will commence with stability levels gradually decreasing from level eight to level four. Each test will last 30 seconds, with patients maintaining the cursor within the smallest balance zones. Postural stability measures will be calculated as the mean of three trials.
medial-lateral stability index | 8 weeks
  It was evaluated using the Biodex Balance System (BBS) before and after the eight-week treatment program. Patients will stand barefoot on the locked platform, centering themselves using visual feedback on the screen. Once stable, foot angles and heel coordinates will be recorded, and tests will commence with stability levels gradually decreasing from level eight to level four. Each test will last 30 seconds, with patients maintaining the cursor within the smallest balance zones. Postural stability measures will be calculated as the mean of three trials.

CONTACTS AND LOCATIONS:
Overall Officials: Haidy Nady Ashem, PhD, Study Chair — Professor, Cairo university
Locations (1):
- Faculty of physical therapy, Cairo University, Giza, Egypt